CLINICAL TRIAL: NCT04233294
Title: Addition of Chidamide to the Combination Treatment of Decitabine Plus Camrelizumab in Combination Treatment Resistant/Relapsed Patients With Classical Hodgkin Lymphoma: an Open-label, Single Arm, Phase II Trial
Brief Title: Addition of Chidamide to the Combination Treatment of Decitabine Plus Camrelizumab in Combination Treatment Resistant/Relapsed Patients With Classical Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-045
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; camrelizumab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chidamide in combination with camrelizumab plus decitabine (Experimental): chidamide 10mg/day, days 1-4, 20mg/day, day 8, 11, 15, 18; camrelizumab 200mg d6; decitabine 10 mg/day, days 1-5, every 3 weeks
  Interventions: Drug: Chidamide; Drug: Camrelizumab; Drug: Decitabine

INTERVENTIONS:
Drug: Chidamide — Chidamide is a novel and orally active benzamide class of HDAC inhibitor that selectively inhibits activity of HDAC1, 2, 3 and 10, which can Induce tumor-cell apoptosis, suppress cell proliferation and enhance immune surveillance.
Drug: Camrelizumab — Camrelizumab is a humanized anti-PD-1 monoclonal antibody.
Drug: Decitabine — Decitabine is an investigational (experimental) drug that works by depleting DNA methyltransferase 1 (DNMT1), which can increase tumor antigens and HLA expression, enhances antigen processing, promotes T cell infiltration, and boosts effector T cell function.

SUMMARY:
This is a Phase II clinical trial for Decitabine plus Camrelizumab resistant/relapsed patients with Hodgkin Lymphoma. The purpose is to evaluate the efficacy and safety of the combination therapy of Chidamide plus Decitabine Plus Camrelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histological confirmation of relapsed or refractory Hodgkin lymphoma (HL).
2. 12 to 75 years of age.
3. ECOG performance of less than 2.
4. Life expectancy of at least 3 months.
5. Subjects with lymphoma must have at least one measureable lesion >1 cm as defined by lymphoma response criteria.
6. Subjects must be relapsed or resistant for the treatment of Decitabine plus Camrelizumab. Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months.
7. Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

1. Subjects with any autoimmune disease or history of syndrome that requires corticosteroids or immunosuppressive medications.
2. Serious uncontrolled medical disorders or active infections, pulmonary infection especially.
3. Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in one month .
4. Prior organ allograft.
5. Women who are pregnant or breastfeeding.
6. Women with a positive pregnancy test on enrollment or prior to investigational product administration.
7. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-02 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  ORR assess by investigators per the 2014 Lugano classification rate of subjects achieved complete response in all evaluable subjects
Adverse effects | 3 years
  Adverse effects were defined according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Nie J, Wang C, Zheng L, Liu Y, Wang C, Chang Y, Hu Y, Guo B, Pan Y, Yang Q, Hu X, Han W. Epigenetic agents plus anti-PD-1 reprogram the tumor microenvironment and restore antitumor efficacy in Hodgkin lymphoma. Blood. 2024 Oct 31;144(18):1936-1950. doi: 10.1182/blood.2024024487. PMID 39093981